CLINICAL TRIAL: NCT07379424
Title: A Single-arm, Phase II, Multi-center Clinical Trial of Sintilimab During the Perioperative Period in Patients With Resectable Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: chen chao Professor (Other)
Responsible Party: Sponsor-Investigator, chen chao Professor, Professor of Clinical, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2025-600(IIT)
Record Dates: First submitted 2025-08-04; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Resectable Locally Advanced Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; Resectable local advanced HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy + PD-1 inhibitor (Experimental): Neoadjuvant therapy: PD-1 inhibitor combined with chemotherapy
  Sintilimab:
  * Specification: 100 mg/10 ml
  * Administration method: 200 mg IV infusion, Q3W, 2 cycles; Standard chemotherapy: paclitaxel (albumin-bound) 260mg/m2 d1+ cisplatin 80mg/m2 d1 or paclitaxel (albumin-bound) 260mg/m2 d1+ nedaplatin 80mg/m2 d1.
  Interventions: Combination Product: Adjuvant therapy: sintilimab combined with radiotherapy

INTERVENTIONS:
Combination Product: Adjuvant therapy: sintilimab combined with radiotherapy — The efficacy was assessed following 2 cycles of neoadjuvant therapy. Patients with efficacy evaluated as CR/PR/SD/PD underwent surgical resection. After surgical resection, sintilimab combined with radiotherapy was initiated as adjuvant therapy, and sintilimab was administered at a dosing interval of Q3W for 15 cycles.

SUMMARY:
This study is a single-arm, multi-center Phase II clinical trial. As depicted in the following study design diagram, its objective is to observe and assess the efficacy and safety of sintilimab during the perioperative period in patients with resectable locally advanced head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
The study aims to recruit patients with head and neck squamous cell carcinoma that has been histologically or cytologically confirmed. The patients should be newly diagnosed, resectable, locally advanced, and have not received any treatment for malignant tumors, as evaluated by the researchers. After signing the informed consent and being screened to meet the inclusion and exclusion criteria, the patients will first receive sintilimab in combination with standard chemotherapy (the specific drugs will be determined by the researchers). Sintilimab will be administered at a dosage of 200 mg, once every three weeks (Q3W).It is administered via intravenous infusion on the first day of each cycle. Efficacy evaluation is conducted after two cycles of treatment. For patients who show a response of complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD) during the efficacy evaluation, surgical resection will be performed. Following surgical resection, sintilimab combined with radiotherapy will be initiated. Sintilimab is administered every three weeks for a total of 15 cycles. Treatment will continue until disease progression, recurrence, intolerable toxicity, withdrawal of informed consent, initiation of other anti-tumor treatments, death, or other circumstances specified in the protocol that necessitate treatment discontinuation, whichever occurs first. The study employs RECIST v1.1 for imaging assessment. The baseline assessment will be conducted within 28 days prior to enrollment. Following 2 cycles of neoadjuvant therapy, a tumor imaging assessment will be performed once. After surgical resection, tumor imaging assessments will be conducted every 3 months (±7 days). If the imaging examination prior to signing the Informed Consent Form (ICF) is within 28 days before the initiation of treatment, it can be utilized as a screening period examination. For subjects who discontinue treatment for reasons other than disease recurrence or death, imaging assessments will also be carried out every 3 months during the first two years after treatment completion, and then every 6 months starting from the third year until a progression or death event occurs. The study will also delve into predictive efficacy biomarkers. For subjects who have signed the informed consent for biomarker sample collection, biomarker blood samples and tumor samples will be collected during the baseline period and throughout the trial. This includes possible tumor biopsies during the baseline period.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent was obtained before any trial-related procedures were performed; 2. Male or female ≥18 years old; 3. Patients with locally advanced squamous cell carcinoma of the head and neck, including oral, oropharyngeal, hypopharyngeal, and laryngeal cancers (except nasopharyngeal and paranasal sinus cancers), confirmed histologically or cytologically by investigator assessment as resectable, including oral, oropharyngeal, hypopharyngeal, and laryngeal cancers; 4. Enrollment stage: stage III-IVA (AJCC 8th); 5. Operable and willing to accept radical surgery after evaluation by multidisciplinary team; 6. The patient had not received any anti-tumor treatment, including but not limited to surgery, radiotherapy, chemotherapy, immunotherapy, targeted therapy, etc.

7. At least one radiographic measurable lesion according to response Evaluation Criteria in Solid Tumors (RECIST, version 1.1); 8. ECOG PS score of 0-1; 9. Expected survival time > 3 months; 10. Adequate organ function, subject must meet the following laboratory indicators:

1. absolute neutrophil count (ANC) ≥1.5x109/L without using granulocyte colony-stimulating factor for the past 14 days.
2. platelet count ≥100×109/L without blood transfusion in the past 14 days.
3. hemoglobin &gt in the absence of blood transfusion or erythropoietin use in the last 14 days; 9g/dL;
4. Total bilirubin ≤1.5× upper limit of normal value (ULN);
5. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN
6. serum creatinine ≤1.5×ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 ml/min;
7. good coagulation function, defined as INR or PT ≤1.5 times ULN;
8. Euthyroid, defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH was beyond the normal range, the subjects could be included if the total T3 (or FT3) and FT4 were within the normal range.
9. Myocardial enzymes within the normal range (simple laboratory abnormalities that were judged by the investigators as not clinically significant were also allowed); 11. For women of childbearing age, a negative urine or serum pregnancy test should be performed within 3 days before receiving the first dose of study drug (day 1 of cycle 1). If a urine pregnancy test result could not be confirmed as negative, a blood pregnancy test was requested. Women who were not of reproductive age were defined as those who had been postmenopausal for at least 1 year or had undergone surgical sterilization or hysterectomy.

12. If there was a risk of pregnancy, all subjects (male or female) were required to use contraception with an annual failure rate of less than 1% throughout the treatment period until 120 days after the last dose of study drug on treatment (or 180 days after the last dose of chemotherapy drug).

Exclusion Criteria:

1. Nasopharyngeal or paranasal sinus cancer;
2. Distant metastasis confirmed by clinical or imaging examination;
3. Malignant diseases other than head and neck squamous cell carcinoma (excluding radical basal cell carcinoma, skin squamous cell carcinoma, and/or radical resection carcinoma in situ) diagnosed within 3 years before the first dose;
4. Currently participating in an interventional clinical study treatment, or receiving another study drug or using a study device within 4 weeks before the first dose;
5. Previous therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or an agent targeting another T-cell receptor that stimulates or coinhibits it (e.g., CTLA-4, OX-40, CD137);
6. Received anti-tumor Chinese patent medicine or immunomodulatory drugs (including thymosin, interferon and interleukin, except for local use to control pleural effusion) with systemic treatment within 2 weeks before the first dose;
7. Active autoimmune disease requiring systemic therapy (e.g., disease-modifying agents, glucocorticoids, or immunosuppressive agents) occurred within 2 years before the first dose. Alternative therapies (e.g., thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency) were not considered systemic therapy;
8. Receiving systemic glucocorticoids (excluding topical glucocorticoids by nasal spray, inhalation, or other route) or any other form of immunosuppressive therapy within 7 days before the first study dose; Note: Physiologic doses of glucocorticoids (prednisone ≤10mg/ day or equivalent) were allowed.
9. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
10. Known to be allergic to sintilimab or excipients;
11. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV1/2 antibody positive);
12. Untreated active hepatitis B (defined as both HBsAg positivity and HBV-DNA copies greater than the upper limit of normal in the laboratory of the participating center);

    Note: Subjects with hepatitis B who met the following criteria were also eligible for inclusion:
    1. HBV viral load &lt before the first dose; 1000 copies /ml (200IU/ml), subjects should receive anti-HBV therapy throughout the study chemotherapy to avoid viral reactivation
    2. Subjects with anti-HBc (+), HBsAg (-), anti-hbs (-), and HBV viral load (-) do not require prophylactic anti-HBV therapy, but close monitoring for viral reactivation is required
13. Active HCV-infected subjects (HCV-antibody positive with an HCV-RNA level above the lower limit of detection);
14. Have received a live vaccine within 30 days before the first dose (cycle 1, day 1); Note: Administration of injectable inactivated virus vaccine against seasonal influenza within 30 days before the first dose is allowed; Live, attenuated, intranasal influenza vaccine was not allowed.
15. Pregnant or lactating women;
16. The presence of any serious or uncontrolled systemic illness, such as:

    1. significant rhythm, conduction or morphological abnormalities on resting ECG that are symptomatic and difficult to control, such as complete left bundle branch block, ≥ Ⅱ degree heart block, ventricular arrhythmia or atrial fibrillation;
    2. unstable angina, congestive heart failure, New York Heart Association (NYHA) class ≥2 chronic heart failure;
    3. any arterial thrombosis, embolism, or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, etc. within 6 months before enrollment;
    4. poor blood pressure control (systolic blood pressure > 140mmHg, diastolic blood pressure > 90mmHg);
    5. a history of noninfectious pneumonia requiring glucocorticoid therapy within 1 year before the first dose or current clinically active interstitial lung disease;
    6. active pulmonary tuberculosis;
    7. presence of active or uncontrolled infection requiring systemic therapy;
    8. clinically active diverticulitis, abdominal abscess, and gastrointestinal obstruction;
    9. liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
    10. poorly controlled diabetes (fasting blood glucose (FBG) > 10mmol/L);
    11. urine routine showed urinary protein ≥++ and confirmed 24-hour urinary protein quantitation > 1.0g;
    12. patients with mental disorders who are unable to cooperate with treatment;
17. Medical history or evidence of disease, treatment or laboratory abnormalities, or other conditions deemed by the investigator to be inappropriate for enrollment that may interfere with the results of the trial or preclude full participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2027-08-25 (Estimated); Study Completion 2028-08-25 (Estimated)

PRIMARY OUTCOMES:
1-year DFS rate | 1 year
  Investigator-assessed relapse-free survival at 1 year according to RECIST v1.1

SECONDARY OUTCOMES:
ORR | Six weeks after enrollment
  The objective response rate was assessed according to RECIST 1.1 criteria
DCR | Six weeks after enrollment
  Disease control rate based on RECIST 1.1 criteria
pCR | Six weeks after enrollment
  Refers to the proportion of patients with no residual tumor in the primary tumor and lymph nodes resected
MPR | Six weeks after enrollment
  Refers to the proportion of patients with ≤10% viable tumor cells in the postoperative resection specimen
OS | Occurrence or end of follow-up（3 years after enrollment), which comes first
  Overall survival
AE | through study completion, an average of 1 year
  The severity of adverse events was graded during the study and during follow-up according to the NCI CTCAE, version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Privacy